CLINICAL TRIAL: NCT07120542
Title: Menopausal Impact on Skin Aging Among Egyptian Women: a Comparative Cross-sectional Study
Brief Title: Menopausal Impact on Skin Aging Among Egyptian Women
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amal Abdulhameed Mostafa, Principal investigator, Sohag University
Other Study IDs: Soh-Med--25-7-1MS
Record Dates: First submitted 2025-07-23; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Skin Aging
MeSH Terms: interventions — Dermoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dermoscopy — dermoscopic assessment of skin aging signs

SUMMARY:
The goal of this study is to understand how menopause affects skin aging in Egyptian women between the ages of 40 and 60.

The main question the study wants to answer is:

Does menopause cause any changes in how the skin ages?

To find out, the participants will be divided into two groups based on their menstrual history:

* Women who have not yet gone through menopause (premenopausal)
* Women who have already gone through menopause (postmenopausal) A researcher will examine the skin of women in both groups to look for signs of aging. Then, the results will be compared to see if there are any differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40 to 60 years
* Egyptian nationality or residency
* Ability to provide informed consent
* Classified as either:

  * Premenopausal (still menstruating regularly)
  * Postmenopausal (no menstruation for ≥12 months)

Exclusion Criteria:

* Menopausal transition (Perimenopausal women
* Menopause induced by hysterectomy
* History of hormone therapy in the past 6 months
* Active dermatological conditions affecting the face (e.g. eczema, psoriasis)
* Use of anti-aging skin treatments (e.g. laser, fillers, retinoids)
* Severe chronic illnesses that may affect skin condition

Ages: 40 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: This study will include Egyptian women between the ages of 40 and 60 years who are either premenopausal or postmenopausal, based on their menstrual history.
  participants must be in good general health and not currently receiving hormone replacement therapy or any treatment known to affect skin condition.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Clinical skin aging severity using Glogau Photoaging Scale | Assessed once at baseline during participant's visit
  The Glogau Photoaging Scale will be used for evaluation. Facial assessment will be conducted both at rest and during facial animation to observe dynamic changes. Participant will be categorized into 4 types or grades where type 1 is mild skin aging and type 4 is severe skin aging
Dermoscopic skin aging score using the dermoscopic photoaging assessment scale | Assessed once at baseline during participant 's visit
  this scale is used to assess facial skin aging. The face will be divided into four regions: the forehead, right cheek, left cheek, and chin. Each region will be examined for the presence of the following features: yellowish discoloration, yellow papules, white linear areas indicating skin atrophy, lentigines, hypo- or hyperpigmented macules, telangiectasia, actinic keratoses, senile comedones, deep wrinkles, superficial wrinkles, and criss-cross wrinkles. Scoring follows a binary (yes/no) approach, where the presence of a given feature in any of the four regions scores one point, yielding a total possible score ranging from 0 to 44. a higher score means worse outcome.

SECONDARY OUTCOMES:
Prevalence of specific clinical and dermoscopic aging features | Recorded during clinical and dermoscopic assessment at baseline
Correlation between menopausal status and severity of skin aging | Assessed once at baseline during participant's visit based on menopausal history and skin aging scores
Correlation between menopausal duration and skin aging | Menopausal duration collected via history at baseline; skin aging assessed at baseline

IPD SHARING:
Plan to Share IPD: Undecided